CLINICAL TRIAL: NCT01902836
Title: Efficacy of Human Dialyzed Leukocytes Extracts in Paediatrics Patients With Moderate Atopic Dermatitis.
Brief Title: Efficacy Study of Dialyzed Leukocytes Extracts to Treat Paediatric Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Polytechnic Institute, Mexico (Other)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, Maria C Jimenez Martinez, PhD, Instituto de Oftalmología Fundación Conde de Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IC-11-06
Record Dates: First submitted 2013-07-11; First posted 2013-07-18 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Childhood Atopic Dermatitis
Keywords: Dialyzable Leukocyte Extracts; Transferon; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Treatment plus DLE (Experimental): Conventional treatment plus DLE
  Conventional treatment: oral Cetirizine 0.25mg/kg, every day, for 4 weeks; chlorpheniramine 0.35 mg/Kg, daily divided in 3 doses, for 4 weeks; and topical Methylprednisolone 0.1% over affected skin area, every 12h for 10 days, then every 24h for 10 days, then every 48h for 10 days and suspend;
  Dialyzed Leukocyte Extracts as Adjuvant Treatment: oral DLE (Transferon) (2mg/5mL), then every day for 5 days, and then every 72hrs to complete one month.
  Interventions: Biological: Conventional treatment plus DLE
- Conventional treatment plus placebo (Placebo Comparator): Conventional treatment plus placebo:
  oral Cetirizine 0.25mg/kg, every day, for 4 weeks; chlorpheniramine 0.35 mg/Kg, daily divided in 3 doses, for 4 weeks; and topical Methylprednisolone 0.1% over affected skin area, every 12h for 10 days, then every 24h for 10 days, then every 48h for 10 days and suspend; plus oral placebo, every day for 5 days, then every 72hrs to complete one month.
  Interventions: Biological: Conventional treatment plus placebo

INTERVENTIONS:
Biological: Conventional treatment plus DLE — Paediatric patients with diagnosis of atopic dermatitis according to Hanifin and Rajka and evaluated with SCORAD as moderate atopic dermatitis were included. Patients were randomized and received in a double blind placebo-controlled treatment:
  Group 1: Conventional treatment plus DLE Conventional Treatment: oral Cetirizine 0.25mg/kg, every day, for 4 weeks; chlorpheniramine 0.35 mg/Kg, daily divided in 3 doses, for 4 weeks; and topical Methylprednisolone 0.1% over affected skin area, every 12h for 10 days, then every 24h for 10 days and then every 48h for 10 days and suspend; plus oral DLE (Transferon) (2mg/5mL), every day for 5 days, then every 72hrs to complete one month
  Other Names: Transferon; Dialyzable Leukocytes Extracts
  Arms: Conventional Treatment plus DLE
Biological: Conventional treatment plus placebo — Group 2: Conventional treatment plus placebo. Conventional treatment: Cetirizine 0.25mg/kg oral, every day, for 4 weeks; chlorpheniramine 0.35 mg/Kg, daily divided in 3 doses, for 4 weeks; topical Methylprednisolone 0.1% over affected skin area, every 12h for 10 days, then every 24h for 10 days and then every 48h for 10 days and suspend; and oral placebo, every day for 5 days, then every 72hrs to complete one month.
  Arms: Conventional treatment plus placebo

SUMMARY:
Patients with atopic dermatitis treated with conventional treatment plus Dialyzed Leukocyte Extracts (DLE-oral Transferon) as adjuvant, have better clinical outcome than patients treated only with conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis diagnosis by Hanifin and Rajka classification
* Dermatitis severity: Moderate, according with SCORAD index.
* Patients without treatment of topical steroids or immunosuppressants in the last 3 weeks.
* Patients with "informed consent form" signed by both parents, or advisor.
* Patients 7 years old or older whom have signed the assent form

Exclusion Criteria:

* Patient who were treated with topical, or systemic steroids and/or immunosuppressants and they cannot discontinue their treatment.
* Patients who lived far from the hospital and they could not go to the visits.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcome evaluated by SCORAD | Day 14
  To determine clinical outcome by SCORAD.

SECONDARY OUTCOMES:
Immunophenotypical changes induced by adjuvant treatment (DLE) (oral Transferon) | 28 days
  To evaluate immunophenotypical changes, on peripheral blood mononuclear cells (PBMC) before, at day 14, and end of treatment.
  Immunophenotypical changes in this study are defined as changes in CLA and CD103 expression on PBMC; and changes in frequency of CD4+CD25+FOXP3 regulatory T cells, before, at day 14, and at end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mirna Toledo, MD, Principal Investigator — Hospital Infantil de Mexico Federico Gomez
Locations (1):
- Hospital Infantil de México, Fedérico Gómez, Mexico City, Mexico City, Mexico